CLINICAL TRIAL: NCT00080106
Title: A Phase II Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Antiretroviral Effect of Immunization With the MRK Ad5 HIV-1 Gag Vaccine in HIV-1 Infected Individuals Who Interrupt Antiretroviral Therapy
Brief Title: Effectiveness of and Immune Response to HIV Vaccination Followed by Treatment Interruption in HIV Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5197; 10014 (Registry Identifier: DAIDS ES); ACTG A5197
Record Dates: First submitted 2004-03-23; First posted 2004-03-25 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2013-07

CONDITIONS: HIV Infections
Keywords: HIV Therapeutic Vaccine; Treatment Experienced; Treatment Interruption; Adenovirus Vector
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Participants in the experimental arm will receive the MRK Ad5 HIV-1 gag vaccine on Day 1, Week 4 and Week 26. Participants will take their antiretroviral medications during the first 3 months of the study.
  Interventions: Biological: MRK Ad5 HIV-1 gag vaccine
- 2 (Placebo Comparator): Participants in Arm 2 will receive a placebo vaccine on Day 1, Week 4 and Week 26. Participants will take their antiretroviral medications during the first 3 months of the study.
  Interventions: Other: Vaccine placebo

INTERVENTIONS:
Biological: MRK Ad5 HIV-1 gag vaccine — MRK Ad5 HIV-1 gag vaccine injected into the upper arm muscle.
  Arms: 1
Other: Vaccine placebo — MRK Ad5 HIV-1 gag placebo vaccine injected into the upper arm muscle.
  Arms: 2

SUMMARY:
HIV vaccines may help the immune systems of HIV infected patients better control the virus. The goal of this study is to determine whether patients on anti-HIV medications can stop taking those medications if they receive an HIV vaccine. While taking anti-HIV medications, participants will receive either an HIV vaccine or a placebo. Participants will then stop taking their anti-HIV medications and the study will compare the viral loads of participants who received the vaccine with the viral loads of participants who received the placebo.

Primary study hypotheses: 1)The Week 12 and Week 16 post-ART interruption geometric mean HIV-1 RNA levels will be lower among participants who had received MRK Ad5 vaccine prior to ART interruption than among participants who received placebo; 2) the time averaged area under the curve of the log10 HIV-1 RNA copies/ml versus day function in the 16 week post-ART interruption step will be lower among participants who received the MRK Ad5 vaccine prior to ART interruption than among participants who receive placebo.

DETAILED DESCRIPTION:
Antiretroviral therapy (ART) has a significant impact on HIV disease; however, HIV cannot be cured with current drug regimens. While the majority of patients initially benefit from ART, drug regimens subsequently fail for many patients due to drug resistance, poor adherence, or toxicity. If given while HIV replication is kept in check by ART, an HIV vaccine may be able to generate an effective long-term immune response capable of controlling the virus, even if ART is discontinued.

The MRK Ad5 HIV-1 gag vaccine uses a replication-defective adenovirus vector and has been found safe in clinical trials of both HIV infected and HIV uninfected adults. This study will evaluate the ability of immunization with the MRK Ad5 HIV-1 gag vaccine to control HIV replication in individuals undergoing treatment interruption. The study will enroll individuals whose HIV replication has been successfully suppressed with ART for at least 2 years.

Participants in this study will be randomly assigned to receive either vaccine or placebo. Both vaccine and placebo will be injected into the upper arm muscle. Participants will take their antiretroviral medications during the first 3 months of the study. Injections will be given on Day 1, Week 4, and Week 26. A study nurse will call participants 1 or 2 days after each injection and participants will be asked to fill out a card with any reactions they have to the injections. About 3 months after the third injection, participants will stop taking their antiretroviral medications for 4 months. Participants will have study visits every 2 to 3 weeks while off medication. After 4 months, participants will have the option of restarting antiretroviral medications or continuing without medication. Participants will then have study visits every 2 months for 8 months. Study visits will include physical exams and blood collection.

All participants will continue to see their primary care provider for HIV treatment and will be restarted on antiretroviral medications if clinically indicated. Participants or their primary care provider will be contacted by phone for updates every 6 months for an additional 3.5 years.

ELIGIBILITY:
Inclusion Criteria

* HIV infected
* On a stable antiretroviral medication regimen (no changes to treatment within 4 weeks of study entry)
* Viral load less than 50 copies/ml
* Viral suppression for 2 years prior to study entry (documented viral loads less than 500 copies/ml)
* CD4 count of 500 cells/mm3 or greater
* Ad5 neutralizing antibody less than 200 units at screening
* Willing to stop antiretroviral medications for at least 16 weeks post-vaccination
* Hepatitis B surface antigen negative
* Weight more than 110 lbs
* Willing to use acceptable methods of contraception

Exclusion Criteria

* Two consecutive viral loads of 500 copies/ml or greater at least 14 days apart during the 24 months prior to study entry
* Two consecutive CD4 counts less than 200 cells/mm3 before starting antiretroviral medications
* History of anaphylaxis
* Allergy to vaccine components
* History of cardiac, pulmonary, gastrointestinal, hepatic, renal, pancreatic, or neurologic disease which, in the opinion of the study official, will compromise study participation
* Pregnancy or breastfeeding
* Contraindication to intramuscular injection, such as anticoagulant therapy or thrombocytopenia
* Immune globulin or blood products within 3 months prior to study entry
* Live vaccine within 30 days prior to study entry
* Inactivated vaccine within 14 days prior to study entry
* Previous HIV vaccine
* History of an AIDS-defining illness. Patients with a history of Kaposi's sarcoma limited to the skin may participate.
* Currently taking drugs or other substances not approved by the FDA. Patients may be on antiretroviral agents not yet approved by the FDA as part of a clinical trial or through an expanded access program.
* Immunomodulatory agents (interferon, IL-2, GM-CSF, systemic corticosteroids, etc.) within 30 days prior to study entry
* Active alcohol or substance abuse which may interfere with the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2004-06; Primary Completion 2007-09 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Analytical treatment interruption (ATI) HIV-1 RNA set-point | Throughout study
ATI log10 HIV-1 RNA copies/ml at all scheduled evaluations during Step II (ATI) | Throughout Step 2

CONTACTS AND LOCATIONS:
Overall Officials: Robert T. Schooley, MD, Study Chair — University of Colorado, Denver
Locations (28):
- United States (27):
  - UCLA CARE Center CRS, Los Angeles, California
  - Stanford CRS, Palo Alto, California
  - Univ. of California Davis Med. Ctr., ACTU, Sacramento, California
  - Ucsd, Avrc Crs, San Diego, California
  - Ucsf Aids Crs, San Francisco, California
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - IHV Baltimore Treatment CRS, Baltimore, Maryland
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - Washington U CRS, St Louis, Missouri
  - Beth Israel Med. Ctr., ACTU, New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Cornell CRS, New York, New York
  - AIDS Care CRS, Rochester, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Case CRS, Cleveland, Ohio
  - MetroHealth CRS, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Pitt CRS, Pittsburgh, Pennsylvania
  - The Miriam Hosp. ACTG CRS, Providence, Rhode Island
  - Univ. of Texas Medical Branch, ACTU, Galveston, Texas
  - University of Washington AIDS CRS, Seattle, Washington
- Puerto Rico-AIDS CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] Shiver JW, Fu TM, Chen L, Casimiro DR, Davies ME, Evans RK, Zhang ZQ, Simon AJ, Trigona WL, Dubey SA, Huang L, Harris VA, Long RS, Liang X, Handt L, Schleif WA, Zhu L, Freed DC, Persaud NV, Guan L, Punt KS, Tang A, Chen M, Wilson KA, Collins KB, Heidecker GJ, Fernandez VR, Perry HC, Joyce JG, Grimm KM, Cook JC, Keller PM, Kresock DS, Mach H, Troutman RD, Isopi LA, Williams DM, Xu Z, Bohannon KE, Volkin DB, Montefiori DC, Miura A, Krivulka GR, Lifton MA, Kuroda MJ, Schmitz JE, Letvin NL, Caulfield MJ, Bett AJ, Youil R, Kaslow DC, Emini EA. Replication-incompetent adenoviral vaccine vector elicits effective anti-immunodeficiency-virus immunity. Nature. 2002 Jan 17;415(6869):331-5. doi: 10.1038/415331a. PMID 11797011
- [Background] Ortiz GM, Wellons M, Brancato J, Vo HT, Zinn RL, Clarkson DE, Van Loon K, Bonhoeffer S, Miralles GD, Montefiori D, Bartlett JA, Nixon DF. Structured antiretroviral treatment interruptions in chronically HIV-1-infected subjects. Proc Natl Acad Sci U S A. 2001 Nov 6;98(23):13288-93. doi: 10.1073/pnas.221452198. Epub 2001 Oct 30. PMID 11687611
- [Background] Moss RB, Brandt C, Giermakowska WK, Savary JR, Theofan G, Zanetti M, Carlo DJ, Wallace MR. HIV-specific immunity during structured antiviral drug treatment interruption. Vaccine. 2003 Mar 7;21(11-12):1066-71. doi: 10.1016/s0264-410x(02)00610-2. PMID 12559781
- [Result] Schooley RT, Spritzler J, Wang H, Lederman MM, Havlir D, Kuritzkes DR, Pollard R, Battaglia C, Robertson M, Mehrotra D, Casimiro D, Cox K, Schock B; AIDS Clinical Trials Group 5197 Study Team. AIDS clinical trials group 5197: a placebo-controlled trial of immunization of HIV-1-infected persons with a replication-deficient adenovirus type 5 vaccine expressing the HIV-1 core protein. J Infect Dis. 2010 Sep 1;202(5):705-16. doi: 10.1086/655468. PMID 20662716
- [Derived] Li JZ, Heisey A, Ahmed H, Wang H, Zheng L, Carrington M, Wrin T, Schooley RT, Lederman MM, Kuritzkes DR; ACTG A5197 Study Team. Relationship of HIV reservoir characteristics with immune status and viral rebound kinetics in an HIV therapeutic vaccine study. AIDS. 2014 Nov 28;28(18):2649-57. doi: 10.1097/QAD.0000000000000478. PMID 25254301
- [Derived] Li JZ, Christensen JA, Wang H, Spritzler J, Kuritzkes DR; AIDS Clinical Trials Group A5197 Study Team. Evaluation of HIV-1 ambiguous nucleotide frequency during antiretroviral treatment interruption. J Acquir Immune Defic Syndr. 2012 Sep 1;61(1):19-22. doi: 10.1097/QAI.0b013e318264460f. PMID 22732468
- [Derived] Li JZ, Brumme CJ, Lederman MM, Brumme ZL, Wang H, Spritzler J, Carrington M, Medvik K, Walker BD, Schooley RT, Kuritzkes DR; AIDS Clinical Trials Group A5197 Study Team. Characteristics and outcomes of initial virologic suppressors during analytic treatment interruption in a therapeutic HIV-1 gag vaccine trial. PLoS One. 2012;7(3):e34134. doi: 10.1371/journal.pone.0034134. Epub 2012 Mar 30. PMID 22479542
- [Derived] Li JZ, Brumme ZL, Brumme CJ, Wang H, Spritzler J, Robertson MN, Lederman MM, Carrington M, Walker BD, Schooley RT, Kuritzkes DR; AIDS Clinical Trials Group A5197 Study Team. Factors associated with viral rebound in HIV-1-infected individuals enrolled in a therapeutic HIV-1 gag vaccine trial. J Infect Dis. 2011 Apr 1;203(7):976-83. doi: 10.1093/infdis/jiq143. PMID 21402549